CLINICAL TRIAL: NCT00047216
Title: A Phase II Study of R115777 (Zarnestra) in Superficial Transitional Cell Carcinoma of Bladder
Brief Title: Tipifarnib in Treating Patients With Recurrent Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-007; CDR0000257564 (Registry Identifier: PDQ (Physician Data Query)); NCI-5612
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer; stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — tipifarnib

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of tipifarnib in treating patients who have recurrent bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 1-year recurrence-free survival rate of patients with stage 0 or I recurrent transitional cell carcinoma of the bladder treated with tipifarnib.

OUTLINE: This is a multicenter study.

Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma (TCC) of the bladder with or without associated carcinoma in situ

  * Stage 0 or I (Ta or T1)
  * Grade 1, 2, or 3 TCC
* Cystoscopically and histologically confirmed recurrent disease after at least 1 course of standard first-line intravesical therapy (e.g., BCG or mitomycin) within the past 12 months
* Complete transurethral resection of bladder tumor performed within past 4 weeks

  * Rendered clinically and cystoscopically tumor free
  * Negative cytology
* No upper tract TCC by intravenous pyelogram, retrograde pyelogram, or CT scan of kidneys (with contrast)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 1 year

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 1.25 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension

Other

* Able to swallow and retain oral medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions to compounds of similar chemical or biological composition to study drug (e.g., other imidazoles such as ketoconazole and other imidazole-based antifungal agents, losartan, metronidazole, or cimetidine)
* No other prior or concurrent malignancy within the past 5 years except nonmelanomatous skin cancer
* No other uncontrolled concurrent illness that would preclude study participation
* No ongoing or active infection
* No active peptic ulcer disease
* No psychiatric illness or social situation that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior systemic chemotherapy for bladder cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for bladder cancer

Surgery

* See Disease Characteristics

Other

* No single-dose post-transurethral resection (TUR) adjuvant intravesical therapy (after TUR that is performed immediately preceding study entry)
* At least 4 weeks since prior investigational agents
* No concurrent commercial or other investigational agents or therapies for malignancy
* No other concurrent therapy for bladder cancer
* No concurrent combination anti-retroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
1-year recurrence-free survival

SECONDARY OUTCOMES:
Recurrence rate at 3, 6, 9, and 12 months
Progression rate at 3, 6, 9, and 12 months
Survival rate
Time to treatment failure
Molecular changes in the host tissue

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chin, MD, Study Chair — London Health Sciences Centre
Locations (7):
- United States (2):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
- Canada (5):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Sunnybrook and Women's College Health Sciences Centre, North York, Ontario
  - Princess Margaret Hospital, Toronto, Ontario